CLINICAL TRIAL: NCT05560516
Title: A Comparison Between Qutenza and Duloxetine for the Treatment of Painful Chemotherapy-induced Peripheral Neuropathy: a Pragmatic Randomized Controlled Trial
Brief Title: Qutenza Versus Duloxetine in Chemotherapy-induced Peripheral Neuropathy (CIPN)
Acronym: QULOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Leiden University Medical Center (Other); Reinier de Graaf Groep (Other)
Responsible Party: Principal Investigator, Emma Cassee, MD, Coordinating investigator/project leader, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL79669.029.21
Record Dates: First submitted 2022-08-15; First posted 2022-09-29 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Qutenza; Duloxetine; Chemotherapy-induced Peripheral Neuropathy; CIPN - Chemotherapy-Induced Peripheral Neuropathy
MeSH Terms: interventions — Capsaicin; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with chemotherapy-induced peripheral neuropathy who receive Qutenza (Experimental)
  Interventions: Drug: Qutenza
- Patients with chemotherapy-induced peripheral neuropathy who receive Duloxetine (Active Comparator)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Qutenza — Capsaicine patch: Qutenza 8% patch will be applied to the skin according to the instruction of the manufacturer. After application of local anesthetics on the skin, a Qutenza 8% patch will be placed. 1-4 patches will be placed and can be adjusted to the right size, depending on the surface of the CIPN. The patch(es) will be removed after 30-60 minutes. The effect will last about 12 weeks.
  Arms: Patients with chemotherapy-induced peripheral neuropathy who receive Qutenza
Drug: Duloxetine — Duloxetine tablets: In week 1 patients will receive 30 mg duloxetine one time per day. In week 2 the dose will be increased to 60 mg one time per day. In case of inacceptable adverse events the patient is allowed to reduce the dose to 30 mg one time per day after consultation with the researcher or physician.
  Arms: Patients with chemotherapy-induced peripheral neuropathy who receive Duloxetine

SUMMARY:
The primary objective is to determine whether in patients with CIPN pain, treatment with Qutenza has the same effect as treatment with duloxetine 60 mg daily.

DETAILED DESCRIPTION:
Rationale: Painful polyneuropathy occurs in approximately 20-40% of patients after the chemotherapy treatment and has a negative influence on quality of life. To our knowledge, no previous randomized study examined Qutenza in patients with CIPN, and no study compared Qutenza to duloxetine. We hypothesize that the effect of Qutenza on the severity of pain and its impact on functioning is the same as that of duloxetine in patients with CIPN, as measured by the numeric rating scale (NRS).

Objective: The primary objective is to determine whether in patients with CIPN pain, treatment with Qutenza has the same effect as treatment with duloxetine 60 mg daily.

Study design: The study is a pragmatic randomized controlled trial.

Study population: Patients who have been treated with chemotherapy in the last 5 years to 3 months and with CIPN grade 1 or higher according to the NCIC-CTC (National Cancer Institute of Canada-Common Toxicity Criteria). The patients are ≥ 18 years of age and have to experience painful neuropathy longer than 3 months with mean (1 week) pain score of ≥4.

Intervention: The affected extremity or extremities will be treated with Qutenza (179mg) according to normal procedures of the hospital and as recommended by the manufacturer.

Patients randomized to duloxetine will start with duloxetine 30 mg per day. After 1 week the dose of duloxetine will be increased, if tolerated, to 60 mg per day for a period of 12 weeks.

Main study parameters/endpoints: The primary endpoint will be average pain reduction at week 12 after start of treatment as measured by the NRS (Numeric Rating Scale). Furthermore secondary objectives will be: pain interference as measured by the BPI (Brief Pain Inventory), side effect profile, quality of life, patient satisfaction, pain at 6 weeks after the start of treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will visit the research location for a screening visit to determine whether the patient fits the in- and exclusion criteria. After the baseline visit patients will be randomized to either receive Qutenza or duloxetine.

All patients will fill in questionnaires (either digital or on paper) before starting treatment with Qutenza or duloxetine (T=0), after 6 weeks of treatment (T=6) and after 12 weeks of treatment (T=12) to obtain the primary and secondary endpoints. All patients will be followed for a total period of 12 weeks. In the first week of treatment patients fill in a questionnaire with side effect profile on a daily basis after 2 weeks patients will fill in a questionnaire on a weekly base. Castor will be used to send the 'side effect questionnaire'.

Since both treatments are commonly used in the treatment of neuropathic pain and are both registered for that indication, no serious complications and no additional burden other than normal treatment are expected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Presence of CIPN grade 1 or higher according to the NCIC-CTC
* Mean pain (1 week) score of ≥ 4
* Treatment with chemotherapy in the last 5 years
* Able to give oral and written informed consent
* Painful neuropathy longer than three months

Exclusion Criteria:

* Peripheral neuropathy from other causes (e.g. carpal/tarsal tunnel syndrome, radiculopathy, spinal stenosis, brachial plexopathy)
* Leptomeningeal carcinomatosis
* Severe depression or use of anti-depressant medication
* Psychiatric disorders which can interfere with cooperation
* Abnormal renal (< GFR 30) or liver function tests (> 2 times normal value)
* Severe heart failure as determined by the cardiologist
* Allergy for duloxetine or capsaicin
* Skin diseases in hands and/or feet, damaged skin
* The presence of uncontrolled/untreated hypertension
* Concomitant use of medication that may interact with duloxetine such as fluvoxamine, ciprofloxacin and enoxacin
* Active cancer treatment (such as radiotherapy or chemotherapy)
* Active cancer
* Previous treatment with Qutenza or duloxetine for CIPN
* Any condition that by the judgement of the investigator might interfere with the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Average pain change | 12 weeks
  As measured by the Brief Pain Inventory, a scale from 0 to 10, with 0 is no pain at all, and 10 is worst pain you can imagine

SECONDARY OUTCOMES:
Pain interference score | 12 weeks
  Measured by the Brief Pain Inventory, a scale from 0 to 10, with 0 is no pain at all, and 10 is worst pain you can imagine
Quality of life score | 12 weeks
  Measured by EuroQol-5D-5L: The descriptive system comprises 5 dimensions: mobility, self care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions
Side effect profile | 12 weeks
  Measured by patient diary, open to fill in what side effects patients experienced
Patient satisfaction | 12 weeks
  Measured by Global perceived effect score, a scale from 1 to 7, with recovery scale 1 means much better and 7 means pain got worse
Pain at 6 weeks after the start of treatment | 6 weeks
  Measured by Brief Pain Inventory, a scale from 0 to 10, with 0 is no pain at all, and 10 is worst pain you can imagine

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, locatie VUMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.2147/jpr.s213912
- See also: Related Info — https://doi.org/10.1097/01.nnr.0000289503.22414.79
- See also: Related Info — https://doi.org/10.1007/s40265-018-0982-7
- See also: Related Info — https://doi.org/10.1016/j.jpainsymman.2020.06.026
- See also: Related Info — https://doi.org/10.2147/jpr.s30406
- See also: Related Info — https://doi.org/10.1007/s00280-018-3664-y
- See also: Related Info — https://www.who.int/data/gho/data/themes/mortality-and-global-health-estimates
- See also: Related Info — https://doi.org/10.1016/j.tox.2011.10.019
- See also: Related Info — https://doi.org/10.3389/fphar.2017.00086
- See also: Related Info — https://doi.org/10.1007/s40261-019-00882-6
- See also: Related Info — https://doi.org/10.1016/j.pain.2014.09.020
- See also: Related Info — https://doi.org/10.1213/01.ane.0000204318.35194.ed
- See also: Related Info — https://www.cancer.gov/about-cancer/treatment/side-effects
- See also: Related Info — https://doi.org/10.1097/md.0000000000018653